CLINICAL TRIAL: NCT05548946
Title: Empirical Evaluation and Clinical Relevance of a Dimensional Model for Personality Disorders in Later Life
Brief Title: A Dimensional Model for Personality Disorders in Later Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Alexianen Zorggroep Tienen (Unknown); Mondriaan (Unknown); GGZ Breburg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BUN:1432021000713
Record Dates: First submitted 2022-09-09; First posted 2022-09-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Psychiatric Disorders
Keywords: Personality Psychology; Aging; Psychological Assessment
MeSH Terms: conditions — Mental Disorders | interventions — Self Report

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General population (Other): In this group, younger adults (18-64) and older (from 65 and older) from the general population are included. The participants fill in questionnaires.
  Interventions: Other: PID-5-BF+M and LPFS-BF 2.0 (self-report questionnaires)
- Clinical Population (Other): In this group, in- and outpatients from the clinical population are included. This are older adults, from the age of 65 with varying psychological pathologies (such as anxiety disorders, mood disorders, substance use disorders, developmental disorders, personality pathology, grief, trauma-related disorders, psychosocial problems, psychosis and schizophrenia-related disorders and somatic disorders). The patients fill in questionnaires and a randomly selected smaller group of patients will conduct a clinical interview.
  Interventions: Other: PID-5-BF+M and LPFS-BF 2.0 (self-report questionnaires); Other: Secondary Questionnaires (self-report and informant questionnaires); Diagnostic Test: Clinical Ratings of the dimensional model; Other: PID-5-BF+M and LPFS-BF 2.0 (Informant questionnaires)

INTERVENTIONS:
Other: PID-5-BF+M and LPFS-BF 2.0 (self-report questionnaires) — All participants will be asked to fill in the PID-5-BF+M and the LPFS-BF 2.0 to examine personality disorders as defined by the AMPD and ICD-11.
  PID-5-BF+M consists of 36 self-report items. It has 18 facet scales and 6 domain scales (Anankastia, Negative Affectivity, Antagonism, Disinhibition, Psychoticism and Detachment).
  The LPFS-BF 2.0 has 12 items, measuring 4 domains of personality functioning (identity, intimacy, self-direction and empathy).
Other: Secondary Questionnaires (self-report and informant questionnaires) — The patients fill in a standard test battery during the first weeks of their admission in the institutions, including questionnaires and interviews. The research team will analyze the results retrospectively.
  This includes:
  YSQ- SF16 (Young & Brown, 1994; Pauwels et al., 2018) GPS (van Alphen et al., 2006) HoNOS 65+ (Burns et al., 1999) HAP 2.0 (Barendse & Thissen, 2006) SCL-90-R (Derogatis, 1983; Dutch version: Arrindell, & Ettema, 1975, 1986, 2005) ADP-IV (Schotte & De Doncker, 1998) CERQ (Garnefski et al., 2007) UCL (Scheurs et al., 1994; 1988) BIS/BAS Scales (Carver & White, 1994) EC Scale of the ATQ (Rothbart et al., 2000) BSI (Derogatis, 1975; Dutch version: Beurs, 2008) SIPP-SF (derived from the SIPP-118; Verheul et al., 2008) SMI (Young et al., 2008) WHO-5 (Dutch version: WHO, 1998) SQ3-SF (Young & Brown, 2005) SCID-5-P (First et al., 2017; Dutch translation: Arntz et al., 2017)
  Arms: Clinical Population
Diagnostic Test: Clinical Ratings of the dimensional model — Clinical ratings of criteria A and B will also be collected. Only a small part of the patients will be selected for this, in order to make the research more feasible. The rater (a clinician or researcher) assesses the patient (in terms of level of personality functioning and personality traits) by means of (structured) clinical interviews. Given clinical ratings of the dimensional criteria are not part of the standard care in either institution, the ratings can be conducted by the doctorandus and Master Thesis students, trained by the doctorandus (in order not to overburden the clinicians).
  The clinical interviews that will be used for the ratings are:
  * The Semigestructureerd Interview voor Persoonlijkheidsfunctioneren DSM-5 (STIP) (Hutsebaut et al., 2014).
  * The Structured Clinical Interview for the DSM-5 (SCID-5-AMPD) (First et al., 2018), only if a Dutch translation is available by the time of this intervention.
  Arms: Clinical Population
Other: PID-5-BF+M and LPFS-BF 2.0 (Informant questionnaires) — In the clinical population, participants will be asked to include an informant (family member, partner, friend, acquaintance), to fill in an informant version of the PID-5-BF+M and LPFS-BF 2.0 questionnaires. It is also possible for the patient to participate in the study without giving permission to include an informant. The informant will be asked to fill in the informant versions of the questionnaires, which contain the exact same items as the self-report versions, adjusted to the third person.
  Arms: Clinical Population

SUMMARY:
Research on personality disorders (PDs) in older adults is currently limited. This is surprising, given that PDs are also common in this age group. Moreover, PDs show high co-morbidity with other disorders (both mental and physical) and often have a negative effect on treatment. With this in mind, the conceptualization, diagnosis and treatment of PDs in older adults represents an important task for mental health care. To this end, problems with the current classification of PDs need to be tackled, as they currently complicate this task. The current DSM-5 (Diagnostic and Statistical Manual, Edition 5) (APA, 2013) categorical PD criteria are mainly based on the living conditions of younger adults and are therefore often not suited for PD diagnosis in older adults. Currently, however, a paradigm shift is taking place from a categorical to a dimensional approach of PDs. The "Alternative Model for Personality Disorders" (AMPD) (APA, 2013) and the approach by ICD-11 (International Classification of Diseases 11th Revision) (WHO, 2019) are examples of new, dimensional models for PDs. These models conceptualize PDs using two dimensional criteria: (1) criterion A, which captures the overall level of personality (dis)functioning and (2) criterion B which describes the PD style by pathological/maladaptive personality traits. This paradigm shift offers the possibility to give the aging context the attention it deserves, by examining the suitability of this new dimensional conceptualization of PD among older adults.

The goal of this research is to examine whether the combined AMPD and ICD-11 dimensional approach is appropriate for use in older adults. This will be done by administering instruments capturing criterion A and B in the general population in younger (18-64) and older (65 and older) adults to evaluate their age-neutrality, as well as in a clinical sample of older (65 and older) adults, to empirically evaluate its clinical relevance in later life.

DETAILED DESCRIPTION:
In the current study, the investigators want to give the ageing context the attention it deserves by examining whether the AMPD and ICD-11 approach is appropriate for use in older adults. This will happen by means of two central objectives, each divided in different research questions.

1. The first central objective is the validation of the AMPD and ICD-11 conceptualization of PDs and its corresponding instruments, in older adults. Even though early research shows promising results for the use of dimensional classification in older adults, both of the questionnaires were originally developed and validated in younger adult samples. Therefore, this research is interested in the examination of the model and its corresponding instruments in older adults. The two instruments that will be used in the study are the Level of Personality Functioning Scale - Brief Version 2.0 (LPFS-BF 2.0) (Weekers et al., 2018) and the Personality Inventory for DSM-5 - Brief Version Modified (PID-5-BF+M) (Bach et al., 2020), which measure criterion A and criterion B, respectively. In this study, the abbreviated version of both questionnaires were chosen, in order not to unnecessarily burden the older participants.

   Firstly, the construct validity of the questionnaires in the general population will be examined. Then, the age-neutrality of the questionnaires (i.e. to what extent younger and older adults having the same degree of personality pathology have the same probability of endorsing related items on the questionnaires) will be investigated. In case non-age-neutral items appear, the investigators will adjust these to obtain age-neutrality. This first research question will occur in the general population. After age neutrality has been demonstrated (possibly after adjustments of the questionnaires), the instrument will be applied in the clinical institutions to evaluate the rest of the research questions. In the clinical population, the construct validity of the questionnaires will be investigated. Construct validity will be evaluated by examining the factor structure of the questionnaires and correlations with other measures of psychopathology (e.g. symptoms of depression and anxiety measured by Brief Symptom Inventory or SCL-90-R). Furthermore, the clinical utility of the questionnaires will be investigated, by examining their ability to distinguish individuals with PDs from those without personality pathology. In addition to research on the psychometric qualities of the questionnaires, the investigators will also validate the AMPD and ICD-11 conceptualization of PDs in two criteria, in older patients by examining the incremental validity of criterion A, above and beyond criterion B. This means the investigators will determine the extent to which criterion A and criterion B can be distinguished from each other and whether they can be differentiated from each other (or in other words do not contain (too much) overlapping information).
2. The second central objective focuses on enhancing general knowledge about the structure and characteristics of PDs in older adults, by positioning PDs in a comprehensive framework of psychopathology, namely the HiTOP model (Hierarchical Taxonomy of Psychopathology) (Kotov et al., 2017). The HiTOP model is an empirical dimensional model that brings together PDs and other clinical disorders in a hierarchical structure, based on their shared transdiagnostic factors. To date, this model has not yet been investigated in older adults (Kotov et al., 2021). With this study, the proposed HiTOP structure will be tested in 65+, in order to gain more insight into the underlying transdiagnostic factors that characterize PDs in older adults, with the ultimate goal of better care and treatment tailored to the older patient.

ELIGIBILITY:
Clinical population (inpatients and outpatients)

Inclusion Criteria:

* ONLY older adults: from the age of 65
* Dutch speaking

Exclusion Criteria (as evaluated by the psychiatrists and psychologists of the participating institutions):

* Severe cognitive impairment (Patients who are admitted because of cognitive impairment will be excluded from the participant pool, other than this the psychiatrists and psychologists of the participating institutions will make an evaluation of the patients' cognitive capacities)
* Acute state of mental impairment which would interfere with the reliability of the patients' responses (for example severe psychosis), as evaluated by the psychiatrists and psychologist of the participating institutions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
PID-5-BF+M questionnaire | Throughout the patient's first weeks of being in in- or outpatient, on average 1 month after admission
  Item scores, scale scores and total scores of the questionnaire
  Items:
  - 38 items (36 original items + 2 additional items)
  Scale scores:
  * 19 personality facets (18 original facet scores + additional facet made up from the additional items) (Emotional Lability, Anxiety, Separation Insecurity, Withdrawal, Anhedonia, Intimacy Avoidance, Manipulativeness, Deceitfulness, Grandiosity, Irresponsibility, Impulsivity, Distractibility, Perfectionism, Rigidity, Orderliness, Unusual Beliefs & Experiences, Eccentricity, Perceptual Dysregulation and Perseveration)
  * 7 personality domains (6 original domains + alternative composition of the Anankastia domain)(Negative Affectivity, Detachment, Antagonism, Disinhibition, Anankastia, Psychoticism and Anankastia by Kerber et al., 2019)
LPFS-BF 2.0 questionnaire | Throughout the patient's first weeks of being in in- or outpatient, on average 1 month after admission
  Item scores, scale scores and total scores of the questionnaire
  Items:
  - 12 items
  Scale scores:
  - 4 domains of personality functioning (identity, intimacy, self-direction and empathy)

SECONDARY OUTCOMES:
The PID-5-BF+M informant version questionnaire | Throughout the patient's first weeks of being in in- or outpatient, on average 1 month after admission
  Scale scores and total scores of the questionnaires.
  The informant versions of the questionnaires consist of the same scales as the self-report versions.
LPFS-BF 2.0 informant version questionnaire | Throughout the patient's first weeks of being in in- or outpatient, on average 1 month after admission
  Scale scores and total scores of the questionnaires.
  The informant versions of the questionnaires consist of the same scales as the self-report versions.
The PID-5-BF+M clinical rating | Throughout the patient's hospitalization and the study completion, on average 1 year after the start of data collection
  The total scores and scale scores of the clinical rating.
  After conducting the clinical ratings with STIP and/or SCID-5-AMPD, the rater gives a clinical rating on criterion B as defined by DSM-5:
  A description of the criterion B domains and each of the facets is given, as well as a possibility for rating, ranging from 0 (not at all descriptive) to 3 (extremely descriptive). These scores then make up the clinical scale scores and total score of The PID-5-BF+M.
LPFS-BF 2.0 clinical rating result | Throughout the patient's hospitalization and the study completion, on average 1 year after the start of data collection
  The total scores and scale scores of the clinical rating.
  After conducting the clinical ratings with STIP and/or SCID-5-AMPD, the rater gives a clinical rating on criterion A defined by DSM-5:
  DSM-5 offers descriptions of the four dimensions of criteria A (identity, self-direction, intimacy and empathy) and asks the rater to give an assessment on a Likert-scale ranging from 0 (healthy) to 4 (severely impaired). These scores then make up the clinical scale scores and total score of the LPFS-BF 2.0.
Secondary measures | Throughout the patient's first weeks of being in in- or outpatient, on average 1 month after admission
  The total scores and scale scores of the questionnaires.
  The scores of the secondary questionnaires will be used to examine validity research questions. A list of these instruments can be found in the section interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Morag Facon, Principal Investigator — Vrije Universiteit Brussel
Locations (2):
- Alexianen Zorggroep Tienen, Tienen, Vlaams-Brabant, Belgium
- Mondriaan, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] APA. Diagnostic and Statistical Manual of Mental Disorders, 5th ed. Washington DC: APA. 2013.
- [Background] World Health Organization. ICD-11: International classification of diseases (11th revision). 2019; Retrieved from https://icd.who.int/.
- [Background] Weekers LC, Hutsebaut J, Kamphuis JH. The Level of Personality Functioning Scale-Brief Form 2.0: Update of a brief instrument for assessing level of personality functioning. Personal Ment Health. 2019 Feb;13(1):3-14. doi: 10.1002/pmh.1434. Epub 2018 Sep 19. PMID 30230242
- [Background] Bach B, Kerber A, Aluja A, Bastiaens T, Keeley JW, Claes L, Fossati A, Gutierrez F, Oliveira SES, Pires R, Riegel KD, Rolland JP, Roskam I, Sellbom M, Somma A, Spanemberg L, Strus W, Thimm JC, Wright AGC, Zimmermann J. International Assessment of DSM-5 and ICD-11 Personality Disorder Traits: Toward a Common Nosology in DSM-5.1. Psychopathology. 2020;53(3-4):179-188. doi: 10.1159/000507589. Epub 2020 May 5. PMID 32369820
- [Background] Kotov R, Krueger RF, Watson D, Achenbach TM, Althoff RR, Bagby RM, Brown TA, Carpenter WT, Caspi A, Clark LA, Eaton NR, Forbes MK, Forbush KT, Goldberg D, Hasin D, Hyman SE, Ivanova MY, Lynam DR, Markon K, Miller JD, Moffitt TE, Morey LC, Mullins-Sweatt SN, Ormel J, Patrick CJ, Regier DA, Rescorla L, Ruggero CJ, Samuel DB, Sellbom M, Simms LJ, Skodol AE, Slade T, South SC, Tackett JL, Waldman ID, Waszczuk MA, Widiger TA, Wright AGC, Zimmerman M. The Hierarchical Taxonomy of Psychopathology (HiTOP): A dimensional alternative to traditional nosologies. J Abnorm Psychol. 2017 May;126(4):454-477. doi: 10.1037/abn0000258. Epub 2017 Mar 23. PMID 28333488
- [Background] Kotov R, Krueger RF, Watson D, Cicero DC, Conway CC, DeYoung CG, Eaton NR, Forbes MK, Hallquist MN, Latzman RD, Mullins-Sweatt SN, Ruggero CJ, Simms LJ, Waldman ID, Waszczuk MA, Wright AGC. The Hierarchical Taxonomy of Psychopathology (HiTOP): A Quantitative Nosology Based on Consensus of Evidence. Annu Rev Clin Psychol. 2021 May 7;17:83-108. doi: 10.1146/annurev-clinpsy-081219-093304. Epub 2021 Feb 12. PMID 33577350
- [Background] Kerber A, Schultze M, Muller S, Ruhling RM, Wright AGC, Spitzer C, Krueger RF, Knaevelsrud C, Zimmermann J. Development of a Short and ICD-11 Compatible Measure for DSM-5 Maladaptive Personality Traits Using Ant Colony Optimization Algorithms. Assessment. 2022 Apr;29(3):467-487. doi: 10.1177/1073191120971848. Epub 2020 Dec 28. PMID 33371717
- [Background] Young JE, Brown G. Young Schema-Questionnaire (2nd ed.). In J. E. Young (Ed.), Cognitive therapy for personality disorders: A schema-focused approach. Sarasota, FL: Professional Resource Press. 1994; Rev. ed., 63- 76.
- [Background] Pauwels E, Dierckx E, Smits D, Janssen R, Claes L. Validation of the Young Schema Questionnaire-Short Form in a Flemish Community Sample. Psychol Belg. 2018 Apr 23;58(1):34-50. doi: 10.5334/pb.406. PMID 30479806
- [Background] van Alphen SP, Engelen GJ, Kuin Y, Hoijtink HJ, Derksen JJ. A preliminary study of the diagnostic accuracy of the Gerontological Personality disorders Scale (GPS). Int J Geriatr Psychiatry. 2006 Sep;21(9):862-8. doi: 10.1002/gps.1572. PMID 16955455
- [Background] Burns A, Beevor A, Lelliott P, Wing J, Blakey A, Orrell M, Mulinga J, Hadden S. Health of the Nation Outcome Scales for elderly people (HoNOS 65+). Br J Psychiatry. 1999 May;174:424-7. doi: 10.1192/bjp.174.5.424. PMID 10616609
- [Background] Barendse HPJ, Thissen AJC. Hetero-Anamnestische Persoonlijkheidsvragenlijst (de HAP): handleiding (HAP en HAP-t 2.0 Versie 2.0). Den Bosch, Netherlands. 2006.
- [Background] Derogatis LR. SCL-90: Administration, Scoring and Procedures Manual-I for the Revised Version and other Instruments of the Psychopathology Rating Scale Series. Baltimore, MD: Johns Hopkins University School of Medicine, Clinical Psychometrics Research Unit. 1983.
- [Background] Arrindell WA, Ettema JHM. Symptom checklist: handleiding bij multidimensionale psychopathologie-indicator. Amsterdam, Nederland: Pearson Assessment and Information B.V.. 1975, 1986, 2005.
- [Background] Schotte CK, de Doncker D, Vankerckhoven C, Vertommen H, Cosyns P. Self-report assessment of the DSM-IV personality disorders. Measurement of trait and distress characteristics: the ADP-IV. Psychol Med. 1998 Sep;28(5):1179-88. doi: 10.1017/s0033291798007041. PMID 9794025
- [Background] Garnefski N, Kraaij V. The Cognitive Emotion Regulation Questionnaire: Psychometric features and prospective relationships with depression and anxiety in adults. European Journal of Psychological Assessment. 2007; 23(3): 141-149. https://doi.org/10.1027/1015-5759.23.3.141.
- [Background] Schreurs, Tellegen, Willige. Coping-lijst. Gedrag. 1984; 12: 101-117.
- [Background] Schreurs, Villige, Tellegen, Brosschot. De Utrechtse coping Lijst: uct-handleiding. Lisse: Swets & Zeitlinger. 1988.
- [Background] Carver, White. Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: The BIS/BAS scales. Journal of Personality and Social Psychology. 1994; 67: 319-333.
- [Background] Rothbart MK, Ahadi SA, Evans DE. Temperament and personality: origins and outcomes. J Pers Soc Psychol. 2000 Jan;78(1):122-35. doi: 10.1037//0022-3514.78.1.122. PMID 10653510
- [Background] Derogatis LR. Brief Symptom Inventory. Clinical Psychometric Research. Baltimore. 1975.
- [Background] De Beurs E. Brief symptom inventory handleiding. Leiden: The Netherlands. PITS B.V.. 2008.
- [Background] Verheul R, Andrea H, Berghout CC, Dolan C, Busschbach JJ, van der Kroft PJ, Bateman AW, Fonagy P. Severity Indices of Personality Problems (SIPP-118): development, factor structure, reliability, and validity. Psychol Assess. 2008 Mar;20(1):23-34. doi: 10.1037/1040-3590.20.1.23. PMID 18315396
- [Background] Young, Arntz, Atkinson, Lobbestael, Weishaar, van Vreeswijk, Klokman. Nederlandse versie The Schema Mode Inventory (SMI). 2008.
- [Background] World Health Organisation. Wellbeing Measures in Primary Health Care/The Depcare Project. WHO Regional Office for Europe: Copenhagen. 1998.
- [Background] Young JE, Brown G. Young Schema Questionnaire - Short Form3 (YSQ-S3). New York, NY: Cognitive Therapy Center. 2005.
- [Background] Hutsebaut J, Berghuis H, De Saeger H, Kaasenbrood A, Ingenhoven T. Semistructured interview for personality functioning DSM-5 (STiP 5.1). The Podium DSM-5 research Group of the Netherlands Centre of Expertise on Personality Disorders. Utrecht: Trimbos Institute. 2014.
- [Background] First, Skodol, Bender, Oldham. Structured Clinical Interview for the DSM-5 Alternative Model for Personality Disorders (SCID-AMPD). American Psychiatric Association. 2018.
- [Background] Marjanovic Z, Struthers CW, Cribbie R, Greenglass ER. The Conscientious Re-sponders Scale. SAGE Open. 2014; 4(3). https://doi.org/10.1177/2158244014545964
- [Background] First, Williams, Benjamin, Smith, Spitzer, Arntz. SCID-5-P : gestructureerd klinisch interview voor DSM-5 persoonlijkheidsstoornissen. American Psychiatric Association. Amsterdam: Boom. 2018.